CLINICAL TRIAL: NCT01987349
Title: Protective Mechanisms Against a Pandemic Respiratory Virus: B- Cell, T-cell, and General Immune Response to Seasonal Influenza Vaccine. Year 1, 2009
Brief Title: T-cell And General Immune Response to Seasonal Influenza Vaccine (SLVP018) - Year 1, 2009
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Cornelia L. Dekker, Professor, Pediatrics, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SU-17219-2009; 2U19AI057229-06 (NIH)
Record Dates: First submitted 2013-10-24; First posted 2013-11-19 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Influenza
Keywords: Influenza vaccines; healthy participants; immunity to influenza; identical twins; fraternal twins; non-twins
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Injections, Intramuscular; FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Group A: age 8-17 yo identical twins (Other): Participants will be randomized to receive either Fluzone® (intramuscular) or FluMist® (intranasal)
  Interventions: Biological: Fluzone® (intramuscular); Biological: FluMist® (intranasal)
- Group B: 18-30 yo identical twins (Other): Participants to receive FluMist® (intranasal)
  Interventions: Biological: FluMist® (intranasal)
- Group C: 18-30 yo fraternal twins (Other): Participants to receive FluMist® (intranasal)
  Interventions: Biological: FluMist® (intranasal)
- Group D: 40-49 yo identical twins (Other): Participants to receive FluMist® (intranasal)
  Interventions: Biological: FluMist® (intranasal)
- Group E: 40-49 yo fraternal twins (Other): Participants to receive FluMist® (intranasal)
  Interventions: Biological: FluMist® (intranasal)
- Group F: 70-100 yo twins (Other): Participants to receive Fluzone® (intramuscular)
  Interventions: Biological: Fluzone® (intramuscular)
- Group G: 70-100 yo non-twins (Other): Participants to receive Fluzone® (intramuscular)
  Interventions: Biological: Fluzone® (intramuscular)

INTERVENTIONS:
Biological: Fluzone® (intramuscular) — Licensed seasonal trivalent inactivated influenza vaccine (IIV3)
  Arms: Group A: age 8-17 yo identical twins; Group F: 70-100 yo twins; Group G: 70-100 yo non-twins
Biological: FluMist® (intranasal) — Licensed trivalent seasonal live attenuated influenza vaccine (LAIV3)
  Arms: Group A: age 8-17 yo identical twins; Group B: 18-30 yo identical twins; Group C: 18-30 yo fraternal twins; Group D: 40-49 yo identical twins; Group E: 40-49 yo fraternal twins

SUMMARY:
This study will compare influenza vaccine responses in monozygotic and dizygotic twins.

DETAILED DESCRIPTION:
The investigators plan to study the response to different influenza vaccines much more broadly and deeply across different age groups and with different vaccine modalities and to probe the influence of genetics on these responses using monozygotic and dizygotic twins.

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise healthy, ambulatory children or adults, ages 8-17 years (identical twin pairs), 18-30 years (identical or fraternal twin pairs), 40-49 years (identical or fraternal twin pairs) or 70-100 years (twin or non-twin adults).
2. Willing to complete the informed consent process.
3. Availability for follow-up for the planned duration of the study at least 28 days after immunization.
4. Acceptable medical history and vital signs.
5. Negative urine pregnancy test for women of childbearing potential
6. If the subject is female and of childbearing potential, she must use an acceptable method of contraception and not become pregnant for the duration of the study. (Acceptable contraception includes implants, injectables, combined oral contraceptives, effective intrauterine devices (IUDs), sexual abstinence, or a vasectomized partner).

Exclusion Criteria:

1. Prior vaccination with TIV or LAIV in Fall 2009
2. Allergy to egg or egg products, or to vaccine components, including gentamicin, gelatin, arginine or MSG (for LAIV only), or thimerosal (TIV multidose vials only).
3. Life-threatening reactions to previous influenza vaccinations
4. Asthma (LAIV groups only)
5. Active systemic or serious concurrent illness, including febrile illness on the day of vaccination
6. History of immune deficiency
7. Known or suspected impairment of immunologic function, including, but not limited to, clinically significant liver disease, diabetes mellitus treated with insulin, moderate to severe renal disease, blood pressure >150/95 at screening, or any other chronic disorder which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
8. Hospitalization in the past year for congestive heart failure or emphysema.
9. Chronic Hepatitis B or C
10. Recent or current use of immunosuppressive medication, including glucocorticoids (corticosteroid nasal sprays are permissible).
11. Subjects in close contact with anyone who has a severely weakened immune system should not receive LAIV.
12. Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia).
13. Autoimmune disease (including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
14. History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
15. Use of any anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin, Plavix, Aggrenox may be acceptable after review by investigator.
16. Receipt of blood or blood products within the past 6 months
17. Medical or psychiatric condition or occupational responsibilities that preclude subject compliance with the protocol
18. Inactivated vaccine 14 days prior to vaccination
19. Live, attenuated vaccine within 60 days of vaccination
20. History of Guillain-Barre Syndrome
21. Pregnant or lactating woman
22. Use of investigational agents within 30 days prior to enrollment
23. Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment
24. Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Ages: 8 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia L Dekker, MD, Principal Investigator — Stanford University; Mark M Davis, PhD, Principal Investigator — Stanford University; Garry Nolan, PhD, Principal Investigator — Stanford University; Ann Arvin, MD, Principal Investigator — Stanford University; Stephen Quake, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horowitz A, Strauss-Albee DM, Leipold M, Kubo J, Nemat-Gorgani N, Dogan OC, Dekker CL, Mackey S, Maecker H, Swan GE, Davis MM, Norman PJ, Guethlein LA, Desai M, Parham P, Blish CA. Genetic and environmental determinants of human NK cell diversity revealed by mass cytometry. Sci Transl Med. 2013 Oct 23;5(208):208ra145. doi: 10.1126/scitranslmed.3006702. PMID 24154599
- [Background] Brodin P, Jojic V, Gao T, Bhattacharya S, Angel CJ, Furman D, Shen-Orr S, Dekker CL, Swan GE, Butte AJ, Maecker HT, Davis MM. Variation in the human immune system is largely driven by non-heritable influences. Cell. 2015 Jan 15;160(1-2):37-47. doi: 10.1016/j.cell.2014.12.020. PMID 25594173
- [Derived] Cheung P, Vallania F, Warsinske HC, Donato M, Schaffert S, Chang SE, Dvorak M, Dekker CL, Davis MM, Utz PJ, Khatri P, Kuo AJ. Single-Cell Chromatin Modification Profiling Reveals Increased Epigenetic Variations with Aging. Cell. 2018 May 31;173(6):1385-1397.e14. doi: 10.1016/j.cell.2018.03.079. Epub 2018 Apr 26. PMID 29706550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Numbers listed in the tables reflect individual twins and not twin pairs.
Groups:
- Group A: Age 8-17 yo Identical Twins: Participants will be randomized to receive Fluzone® (intramuscular)
- Group A: Age 8-17yo Identical Twins: Participants will be randomized to receive FluMist® (intranasal)
- Group B: Age 18-30 yo Identical Twins; Group C: Age 18-30 yo Fraternal Twins; Group D: Age 40-49 yo Identical Twins; Group E: Age 40-49 yo Fraternal Twins: Participants to receive FluMist® (intranasal)
- Group F: 70-100 yo Identical Twins; Group G: 70-100 yo Nontwins: Participants to receive Fluzone® (intramuscular)
Period: Overall Study
Arm/Group | Group A: Age 8-17 yo Identical Twins | Group A: Age 8-17yo Identical Twins | Group B: Age 18-30 yo Identical Twins | Group C: Age 18-30 yo Fraternal Twins | Group D: Age 40-49 yo Identical Twins | Group E: Age 40-49 yo Fraternal Twins | Group F: 70-100 yo Identical Twins | Group G: 70-100 yo Nontwins
Started | 6 | 6 | 8 | 6 | 6 | 6 | 10 | 25
Completed | 6 | 6 | 8 | 6 | 6 | 6 | 10 | 24
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants between the ages of 8 - 100 years old.
Groups:
- Group A: Age 8-17 yo Identical Twins (Fluzone): Participants will be randomized to receive Fluzone® (intramuscular)
- Group A: Age 8-17 yo Identical Twins (FluMist): Participants will be randomized to receive FluMist® (intranasal)
- Total: Total of all reporting groups
Arm/Group | Group A: Age 8-17 yo Identical Twins (Fluzone) | Group A: Age 8-17 yo Identical Twins (FluMist) | Group B: Age 18-30 yo Identical Twins | Group C: Age 18-30 yo Fraternal Twins | Group D: Age 40-49 yo Identical Twins | Group E: Age 40-49 yo Fraternal Twins | Group F: 70-100 yo Identical Twins | Group G: 70-100 yo Nontwins | Total
Number analyzed (Participants) | 6 | 6 | 8 | 6 | 6 | 6 | 10 | 24 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 12
  Between 18 and 65 years | 0 | 0 | 8 | 6 | 6 | 6 | 0 | 0 | 26
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 24 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4 | 4 | 4 | 4 | 4 | 18 | 42
  Male | 4 | 4 | 4 | 2 | 2 | 2 | 6 | 6 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 4
  Not Hispanic or Latino | 6 | 6 | 6 | 4 | 6 | 6 | 10 | 24 | 68
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
  White | 6 | 6 | 6 | 6 | 6 | 2 | 10 | 23 | 65
  More than one race | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants From Each Arm Who Received Influenza Vaccine Vaccine
Time Frame: Day 0 to 28
Measure: Count of Participants; unit: Participants
Groups:
- Group A: Age 8-17 yo Identical Twins (IM): Participants will be randomized to receive Fluzone® (intramuscular)
  Fluzone® (intramuscular): Licensed seasonal trivalent inactivated influenza vaccine (IIV3)
- Group A: Age 8-17 yo Identical Twins (IN): Participants will be randomized to receive FluMist® (intranasal
  FluMist®: Licensed trivalent seasonal live attenuated influenza vaccine (LAIV3)
Arm/Group | Group A: Age 8-17 yo Identical Twins (IM) | Group A: Age 8-17 yo Identical Twins (IN) | Group B: 18-30 yo Identical Twins | Group C: 18-30 yo Fraternal Twins | Group D: 40-49 yo Identical Twins | Group E: 40-49 yo Fraternal Twins | Group F: 70-100 yo Twins | Group G: 70-100 yo Non-twins
Number analyzed (Participants) | 6 | 6 | 8 | 6 | 6 | 6 | 10 | 24
Participants | 6 | 6 | 8 | 6 | 6 | 6 | 10 | 24

2. Secondary Outcome: Number of Participants With Related Adverse Events
Time Frame: Day 0 to 28 post-immunization
Measure: Count of Participants; unit: Participants
Groups:
- Group A: Age 8-17 yo Identical Twins (IN): Participants will be randomized to receive FluMist® (intranasal)
  FluMist® (intranasal): Licensed trivalent seasonal live attenuated influenza vaccine (LAIV3)
Arm/Group | Group A: Age 8-17 yo Identical Twins (IM) | Group A: Age 8-17 yo Identical Twins (IN) | Group B: 18-30 yo Identical Twins | Group C: 18-30 yo Fraternal Twins | Group D: 40-49 yo Identical Twins | Group E: 40-49 yo Fraternal Twins | Group F: 70-100 yo Twins | Group G: 70-100 yo Non-twins
Number analyzed (Participants) | 6 | 6 | 8 | 6 | 6 | 6 | 10 | 24
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Other Pre Specified Outcome: Lymphocyte Response to Influenza Immunization
Description: Compare lymphocyte responses at Days 6-14 and the lymphocyte and serology responses at Day 28 post-immunization following annual administration of the influenza vaccines
Time Frame: Day 6-28 post-immunization
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Day 0 to Day 28 of study participation
Description: Clinical Assessment performed at each visit
Groups:
- Group B: 18-30 yo Identical Twin Pairs; Group C: 18-30 yo Fraternal Twins; Group D: 40-49 yo Identical Twins; Group E: 40-49 yo Fraternal Twins: Participants to receive Flumist® (intranasal)
  Flumist® (intranasal): Licensed trivalent seasonal live attenuated influenza vaccine (LAIV3)
Arm/Group | Group A: Age 8-17 yo Identical Twins (Fluzone) | Group A: Age 8-17 yo Identical Twins (Flumist) | Group B: 18-30 yo Identical Twin Pairs | Group C: 18-30 yo Fraternal Twins | Group D: 40-49 yo Identical Twins | Group E: 40-49 yo Fraternal Twins | Group F: 70-100 yo Twins | Group G: 70-100 yo Non-twins
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/8 | 0/6 | 0/6 | 0/6 | 0/10 | 0/24
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/8 | 0/6 | 0/6 | 0/6 | 0/10 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No